CLINICAL TRIAL: NCT01507142
Title: Rapid Oral Test for Therapeutic Response in HIV/AIDS Patients
Status: Completed | Type: Observational
Sponsor: Gaia Medical Institute (Industry)
Collaborators: AIDS Healthcare Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: GAIA-AIDS-001
Record Dates: First submitted 2012-01-06; First posted 2012-01-10 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: AIDS/HIV PROBLEM
Keywords: saliva; diagnostics; HIV; AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- cART-unresponsive AIDS: HIV-positive, AIDS diagnosis, cART for >18 months, <200 CD4 Tcells/mm3 and Viral Load >5000 copies/ml
- cART-responsive AIDS: HIV-positive, AIDS diagnosis, cART for >18 months, >350 CD4 Tcells/mm3 and Viral Load<50 copies/ml
- Acute or early HIV infection: Acute HIV: Acute retroviral syndrome, Negative or positive HIV antibody, Positive HIV p24gag, viral load or NAAT / Early HIV: HIV antibody and viral load positive currently, negative in last 12 months, No clinical or immunological evidence of advanced HIV disease
- HIV-negative Hepatitis B: Negative HIV antibody and viral load, Positive HBV antibody, Positive or Negative HBV surface antigen, Negative or Positive HBV viral load

SUMMARY:
This study has been designed to evaluate a new oral test for therapeutic monitoring of HIV/AIDS patients that are receiving the combination Anti-Retroviral Therapy (cART). The test will measure saliva-based Stress Response Profiling(SRP) biomarkers using laboratory assays. Results of the test will show if HIV/AIDS patients successfully responded to cART. Preliminary studies showed that SRP biomarkers were strongly increased in cART-unresponsive AIDS patients. However, the diagnostic accuracy of the oral test, patients will be recruited to donate saliva: AIDS patients responsive or unresponsive to cART, and controls (acute or early HIV patients, and HIV-negative patients with hepatitis).

The saliva samples will be used to measure SRP biomarker concentrations. Results will show whether the biomarker measurements provide accurate and specific diagnostics for ART response.

ELIGIBILITY:
Inclusion Criteria:

Group 1, cART-unresponsive

* Documented HIV-positive before obtaining AIDS diagnosis
* cART for 18 months or longer
* consistent lab tests in previous 3-6 months: < or equal to 200 CD4 T cells/mm3, viral load >5000 HIV RNA copies/ml

Group 2, cART-responsive

* Documented HIV-positive before obtaining AIDS diagnosis
* cART for 18 months or longer
* consistent lab tests in previous 3-6 months: > or equal to 350 CD4 T cells/mm3, viral load < or equal to 50 HIV RNA copies/ml

Group 3, acute/early HIV

Acute HIV:

* Signs and symptoms of acute retroviral syndrome in a person with either a negative or evolving antibody response (western blot or ELISA) in presence of a positive HIV p24gag antigen or HIV-1 proviral DNA PCR or positive HIV-1 RNA

Early HIV:

* A positive antibody response (western blot or ELISA) with a documented negative serological test or plasma HIV-1 RNA within the past 12 months or a positive ELISA and a negative de-tuned ELISA within 30 days of a positive ELISA specimen in an untreated person with no clinical or immunological evidence of advanced HIV disease (CD4 count >200 cells/mm3 or >14%)

Group 4, HIV-negative Hepatitis-positive

* HIV test negative (western blot, ELISA or viral load)
* Positive Hepatitis B surface antigen and detectable hepatitis B viral load (HCV B RNA), treated or not OR Positive Hepatitis C antibodies and detectable hepatitis C viral load (HCV C RNA), treated or not

Exclusion Criteria:

* Pregnant or lactating women
* Non-adherent patients
* Any conditions which will affect saliva production: e.g. Sjogren's syndrome or chronic mouth dryness
* Cytotoxic chemotherapy, interferon treatment, or radiation therapy within the preceding 3 weeks
* Active alcohol or substance abuse (narcotics or other controlled substances) within 6 months prior to the saliva sampling
* Significant psychiatric illness that in the opinion of the principle investigator might interfere with making an informed decision
* Incapable to give informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HIV-positive, or HIV-negative and Hepatitis-positive adult participants
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2012-09 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Chen, M.D., Principal Investigator — AIDS Healthcare Foundation; Sarka Southern, Ph.D., Principal Investigator — Gaia Medical Institute
Locations (1):
- AIDS Healthcare Foundation, Los Angeles, California, United States